CLINICAL TRIAL: NCT06662630
Title: Assessing the Physiological Impact and Safety of Continuous High-Frequency Oscillatory Ventilation in Critically Ill Patients Under Mechanical Ventilation
Brief Title: Physiological Effects and Safety of Continuous High-frequency Oscillatory Ventilation in Mechanical Ventilation Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZSZZ202410
Record Dates: First submitted 2024-10-19; First posted 2024-10-29 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-10

CONDITIONS: Atelectasis; Acute Respiratory Distress Syndrome; VAP - Ventilator Associated Pneumonia
Keywords: mechanical ventilation; HFOV; EIT; FRC
MeSH Terms: conditions — Pulmonary Atelectasis; Respiratory Distress Syndrome; Pneumonia, Ventilator-Associated

STUDY DESIGN:
Intervention Model Description: Interventional study evaluating the beneficial impact of continuous high-frequency oscillatory ventilation in patients with mechanical ventilation
Masking Description: Analysis of data will be conducted by a statistician not involved in interventions at bedside
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHFO group (Experimental): After checking the availability of the CHFO machine (MetaNeb® system), the inclusion and non-inclusion criteria, the patient is included. The following procedures are performed:
  1. installation of an EIT belt in the 4th or 5th intercostal space (Pulmovista® 500, Dräger)
  2. continuous recording of digital and analogic data After collecting initial data from the patient within 30 minutes before CHFO treatment, successive 10-minutes CHFO were performed. At the end of the treatment, all the data is collected.
  Interventions: Device: High-Frequency Oscillatory Ventilation

INTERVENTIONS:
Device: High-Frequency Oscillatory Ventilation — Administer 10 minutes of high-frequency oscillatory ventilation in mechanically ventilated patients.

SUMMARY:
Mechanical ventilation is an important treatment modality for intensive care unit (ICU) patients, but it also brings a series of problems such as ventilator-associated pneumonia, ventilator-induced lung injury, and atelectasis. Continuous High-Frequency Oscillation (CHFO )is often considered to have a protective effect on the lungs. CHFO provides effective gas exchange at supraphysiological frequencies while minimizing pressure fluctuations, producing tidal volumes smaller than dead space and adjusting around a continuously expanding pressure to optimize end-expiratory lung volume (EELV) by achieving and maintaining lung recruitment. However, the physiological effects and safety of CHFO in critically ill patients on mechanical ventilation lack relevant research. The objective of this research is to assess the feasibility, safety, and efficacy of CHFO in a population of mechanically ventilated critically ill patients.

DETAILED DESCRIPTION:
This is an interventional study evaluating the beneficial impact of CHFO of patients with mechanical ventilation on pathophysiological parameters.

This therapeutic study aims to treat patients using CHFO machine (MetaNeb system). The study consists of comparing pulmonary pathophysiological parameters before and after the treatment of CHFO in patients with invasive mechanical ventilation.

The primary outcome is the difference between the end-expiratory lung volume (EELV) and chest electrical impedance tomography (EIT) measured at the end of CHFO (10 min) and the basal value measured at the beginning of the protocol.

The minimum number of subjects to enroll in this study is 30 patients with invasive mechanical ventilation. Intermediate analyses are planned every 5 patients in order to reevaluate the needed number of patients.

The basal value at the beginning of the protocol, collection of ventilatory parameters on the ventilator, collection of arterial blood gas analyses and measurement of heart rate, and blood pressure. In the middle of treatment, collection of arterial blood gas analyses and measurement of heart rate, and blood pressure. At the end of the treatment, collection of ventilatory parameters on the ventilator, collection of arterial blood gas analyses and measurement of heart rate, and blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 and younger than 90 years;
* Admitted to the ICU after October 15, 2024, who are intubated and expected to be unable to be extubated within 48 hours due to ARDS, or have atelectasis, or have VAP.
* Signed informed consent for MetaNeb treatment.

Exclusion Criteria:

* Refusal to participate in the proposed study.
* Age < 20 years;
* Pregnancy;
* Significant hemodynamic instability defined as an increase of more than 20% in catecholamine doses in the last hour, despite optimization of blood volume, for a target mean blood pressure between 65 and 75 mmHg.
* Participation in another trial within 30 days prior to meeting eligibility criteria;
* Severe chronic respiratory disease requiring long-term oxygen therapy or home mechanical ventilation;
* Pneumothorax;
* Expected duration of mechanical ventilation < 48 hours
* Decision to refuse life-sustaining treatment.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-11-19 (Estimated); Primary Completion 2025-10-14 (Estimated); Study Completion 2026-10-14 (Estimated)

PRIMARY OUTCOMES:
EELV | Baseline, and at the end of intervention (30th minute)
  EELV was measured utilizing the nitrogen washout-washin technique (E-sCOVX module sensor, GE Healthcare, Madison, WI, USA). The infusion of intravenous anesthetic agents and rocuronium bromide was administered to establish controlled mechanical ventilation during EELV measurement. Consistency in ventilator parameters was maintained throughout the EELV monitoring including follow-up measurements. Measurements will be taken at two time points: (1) Within 30 minutes before the start of CHFO and (2) within 30 minutes after its completion.
EIT | Baseline, and at the end of intervention (30th minute)
  In EIT monitoring, a 16-electrode belt was placed around the chest to record signals. Measurements will be taken at two time points: (1) Within 30 minutes before the start of CHFO and (2) within 30 minutes after its completion.

SECONDARY OUTCOMES:
Central venous pressure before and after the CHOF treatment | Baseline, and at the end of the intervention (30 minutes post-intervention)
  The CVC is inserted via the internal jugular vein, subclavian vein, or femoral vein, depending on the patient and their condition. CVP is measured using a pressure measurement system, according to the measurement requirements. Measurements will be taken at two time points: (1) Within 30 minutes before the start of CHFO and (2) within 30 minutes after its completion.
PaO2/FiO2 ratio before and after the CHOF treatment | Baseline, and at the end of the intervention (30 minutes post-intervention)
  The PaO2/FiO2 ratio will be calculated by dividing the partial pressure of arterial oxygen (PaO2) by the fraction of inspired oxygen (FiO2). Measurements will be taken at two time points: (1) Within 30 minutes before the start of CHFO and (2) within 30 minutes after its completion.
Plateau pressure | Baseline, and at the end of the intervention (30 minutes post-intervention)
  Measured during an end-inspiratory pause of 3 seconds.
Mean arterial pressure | Baseline, during intervention, and at the end of intervention (30th minute)
  Mean arterial pressure measured continuously from the radial artery within 30 minutes before and after the treatment of CHOF and during the CHOF treatments.
Adverse events | Baseline, during intervention, and at the end of intervention (30th minute)
  The occurrence of adverse events and the corresponding rate.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Zhou, PhD, Study Director — Fudan University
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China